CLINICAL TRIAL: NCT01582165
Title: Microvascular Resistance in Women With Chest Pain and no or Minimal Coronary Artery Disease
Brief Title: Women With Chest Pain and no Significant Coronary Artery Stenosis; A Study on Microvascular Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Ole Geir Solberg, Consultant, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3tcAZ; 2011-002630-39 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Angina. IMR. Statin. (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Angina. IMR. Placebo. (Placebo Comparator)
  Interventions: Drug: Placebo.

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20 mg once daily vs placebo for 6 months
  Arms: Angina. IMR. Statin.
Drug: Placebo. — Placebo once daily vs rosuvastatin for 6 months
  Arms: Angina. IMR. Placebo.

SUMMARY:
Female patients presenting with persistent chest pain despite no obstructive coronary artery disease have impaired prognosis. Stress tests are often positive or inconclusive. As much as 20% of women with chest pain and minimal angiographic CAD have evidence of myocardial ischemia, suggesting impaired coronary microcirculation. The index of microvascular resistance (IMR) is a method for indirectly investigating microvascular function in the cardiac catheterization laboratory.

66 female patients, age 30-70 years, with chest pain and "normal" or near normal coronary angiograms will be included. After coronary physiologic evaluation, patients will be randomized in a double blind study to rosuvastatin 20 mg/day or matching placebo tablets for altogether 6 months.

The investigators hypothesize that:

1. A substantial number of women with chest pain and normal or minimal pathology on angiograms have microvascular dysfunction defined by a raised IMR.
2. Statins, based on its pleiotropic action will improve endothelial function and thereby IMR.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age 30 - 70 years
3. Chest pain suggestive of symptomatic coronary artery disease
4. A coronary angiogram with no or minimal coronary artery disease
5. Fractional flow reserve value over 0,80

Exclusion Criteria:

1. Male gender
2. Age under 30 years or over 70
3. Coronary artery stenosis ≥ 33 % in any epicardial vessel
4. Fractional flow reserve value ≤ 0,80
5. Pregnant or nursing women
6. Women of childbearing potential not using contraception
7. Short life expectancy
8. Uncontrolled endocrinological disease
9. Arterial hypertension
10. Structural heart disease
11. Significant mental disorder, including dementia
12. Inability to comply with the protocol -

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Temporal changes in microvascular perfusion indices (Index of Microvascular Function (IMR) and Coronary Flow Reserve (CFR)). | 6 months
  During a left heart catheterization IMR and CFR are measured at baseline and at 6 months. Patients are randomized to rosuvastatin vs placebo. The objectives are to determine whether women with chest pain with no or minimal angiographic coronary artery disease, have a raised index of microvascular resistance and to determine whether high-dose statin treatment will modify microvascular perfusion indices in these patients.

SECONDARY OUTCOMES:
Angina pectoris classification (CCS). | 6 months
  Women with chest pain are randomized to rosuvastatin vs placebo. Angina pectoris (CCS classification) will be compared in the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Aaberge, MD, PhD, Principal Investigator — Oslo University Hospital Rikshospitalet, Oslo, Norway
Locations (1):
- Oslo University Hospital, Dep of Cardiology, Rikshospitalet, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Analyses of the study will start within a few weeks or months. Publication planned in 2017

REFERENCES:
- [Derived] Solberg OG, Stavem K, Ragnarsson A, Beitnes JO, Skardal R, Seljeflot I, Ueland T, Aukrust P, Gullestad L, Aaberge L. Index of microvascular resistance to assess the effect of rosuvastatin on microvascular function in women with chest pain and no obstructive coronary artery disease: A double-blind randomized study. Catheter Cardiovasc Interv. 2019 Nov 1;94(5):660-668. doi: 10.1002/ccd.28157. Epub 2019 Feb 21. PMID 30790446